CLINICAL TRIAL: NCT06101797
Title: Remote and In-person Supervised Exercise in Patients With Knee Osteoarthritis (RISE-KOA): a Single Blinded, Randomized, Non-inferiority Trial.
Brief Title: Remote and In-person Supervised Exercise in Patients With Knee Osteoarthritis
Acronym: RISE-KOA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Cristine Lima Alberton, Principal Investigator, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 74411723.0.0000.5313
Record Dates: First submitted 2023-10-16; First posted 2023-10-26 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-02

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: This study is a non-inferiority randomized clinical trial with two parallel groups in a single center with blinding of outcome assessors. Patients, males, and females with symptomatic and radiographic knee OA will be allocated to supervised in-person or remote exercise groups based on a stratified randomization method, considering the baseline outcome age (in the categories of participants aged 45 to 54 years old or 55 to 80 years old). A single independent researcher assistant will carry out randomization with a 1:1 ratio.
Who Masked: Outcomes Assessor
Masking Description: Blinding will be implemented by the outcome assessor. All measurements (PROMs, muscle architecture, and functional outcomes) will be conducted by an evaluator blinded to the participant's group. Due to the nature of the intervention, investigators conducting the exercise intervention and participants will not be able to be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remote supervised exercise group (Experimental): The intervention will last 12 weeks and consist of muscle-strengthening exercises for the lower extremities supervised remotely by video call.
  Interventions: Other: Remote supervised exercise group
- In-person supervised exercise group (Experimental): The intervention will last 12 weeks and consist of muscle-strengthening exercises for the lower extremities supervised in person at a physiotherapy clinic.
  Interventions: Other: In-person supervised exercise group

INTERVENTIONS:
Other: Remote supervised exercise group — The exercise protocol for this group consists of individualized muscle-strengthening exercises for the lower extremities supervised by video call. The intervention will occur 2-3 times per week, each lasting approximately 40 minutes. The exercise protocol will consist of six muscle-strengthening exercises for the lower extremities, which will be guided, alternating muscle groups. In the first two weeks of treatment, exercise intensity will be monitored for participants to complete two sets of 8-12 repetitions in dynamic exercises. From the third week onward, participants will progress to one additional set. Adjustments to weight-bearing, the external load imposed by the elastic band, and exercise position throughout the protocol will be performed to maintain the participant's level of effort. After supervised exercise treatment, patients will be encouraged to maintain an exercise routine with the same exercise protocol, however, without physiotherapy supervision.
  Arms: Remote supervised exercise group
Other: In-person supervised exercise group — The exercise protocol for this group consists of individualized muscle-strengthening exercises for the lower extremities supervised at a physiotherapy clinic. The intervention will occur 2-3 times per week, each lasting approximately 40 minutes. The exercise protocol will consist of six muscle-strengthening exercises for the lower extremities, which will be guided, alternating muscle groups. In the first two weeks of treatment, exercise intensity will be monitored for participants to complete two sets of 8-12 repetitions in dynamic exercises. From the third week onward, participants will progress to one additional set. Adjustments to weight-bearing, the external load imposed by the elastic band, and exercise position throughout the protocol will be performed to maintain the participant's level of effort. After supervised exercise treatment, patients will be encouraged to maintain an exercise routine with the same exercise protocol, however, without physiotherapy supervision.
  Arms: In-person supervised exercise group

SUMMARY:
Exercise supervision via telehealth resources is an alternative to the in-person modality with similar therapeutic effectiveness across different clinical profiles. Especially in the context of knee osteoarthritis (OA), exercise is recommended by international guidelines. However, it is necessary to elucidate the comparability of remote and in-person supervised exercise effectiveness for these patients. Therefore, the study's objective is to investigate the responses of a remote compared to the in-person supervised exercise program on patient-reported outcomes measures (PROMs), muscular architecture, and the functional performance of patients with knee OA. Forty-eight patients with symptomatic and radiographic knee OA will be randomly assigned to remote or in-person exercise programs. The intervention will last 12 weeks, encompassing muscle-strengthening exercises for the lower extremities, with a frequency of twice a week for the initial two weeks and three sessions per week from the third week onwards. Supervision will be conducted remotely via video calls in one group, while the other will receive in-person supervision at a physiotherapy clinic. Program sessions will comprise six exercises. In the first session treatment block, exercises will be guided for the muscle groups of the knee extensors, hip adductors, and plantar flexors, and in the second block, for knee extensors, hip abductors, and knee flexors. After the 12-week supervised treatment period, participants will be encouraged to continue the same exercise program at home without a physiotherapist in the following six weeks. PROMs related to the joint condition will be measured, such as pain, symptoms, daily activities, sports and leisure activities, and quality of life. The psychological domain will also be evaluated, including pain catastrophizing, symptoms of depression, anxiety and stress, and sleep quality. Additionally, measurements of the muscular architecture of the quadriceps femoris, including muscle thickness, pennation angle, fascicle length, and echo intensity, will be taken. Functional performance will be assessed through tests that include the skills of standing and sitting, walking and going up, and down stairs. PROMs will be measured at weeks 0, 6, 12, and 18. Muscular architecture and functional parameters will be measured at weeks 0 and 12. Data analysis will be conducted using Linear Mixed Models, and analysis will be presented by intention to treat and per protocol. The significance level adopted for this study will be α = 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a radiographic diagnosis of unilateral or bilateral knee OA and classified as grades II or III according to the Kellgren and Lawrence criteria (KELLGREN e LAWRENCE, 1957).
* Symptomatic patients according to following American College of Rheumatology criteria - average pain score ≥3 in the last week on the numerical rating scale (0-10), morning stiffness <30 minutes and joint crepitus (ALTMAN et al., 1986).
* Independent walking and internet access.

Exclusion Criteria:

* Patients with systemic inflammatory diseases, including rheumatoid arthritis, ankylosing spondylitis, and systemic lupus erythematosus.
* Neurological diseases with motor disability.
* Unstable heart diseases.
* History of total knee arthroplasty or lower extremity surgery.
* Body mass index (BMI) ≥ 35 kg/m².
* Physical therapy treatment or participation in a supervised exercise program in the last six months.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-03-08 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Baseline (week 0), During intervention (week 6), Post-intervention (week 12).
  Average pain intensity in the last week will be assessed using an 11-point Pain Intensity Numerical Rating Scale (NRS), in which 0 corresponds to "no pain," and 10 represents "worst possible pain." NRS is a patient-reported outcome measure for assessment and clinical decision-making in patients with knee OA with good psychometric properties (ORNETTI et al., 2011).
Physical function | Baseline (week 0), During intervention (week 6), Post-intervention (week 12).
  Physical function will be measured by Knee Injury and Osteoarthritis Outcome Score (KOOS) using an Activities of Daily Living subscale. The KOOS is a patient-reported outcome measure composed of 42 items divided into five subscales: Pain, other Symptoms, Activities of daily living, Sport and Recreation Function, and Knee-related Quality of Life. Its score ranges from 0 (extreme problem) to 100 (no problems) separately in each subscale (COLLINS et al., 2011). The Brazilian version of the KOOS questionnaire was recently validated, consisting of an instrument with validity, reliability, and responsiveness in patients with knee OA (ALMEIDA et al., 2022).

SECONDARY OUTCOMES:
Pain intensity | Follow up period (week 18).
  Average pain intensity in the last week will be assessed using an 11-point Pain Intensity Numerical Rating Scale (NRS), in which 0 corresponds to "no pain," and 10 represents "worst possible pain." NRS is a patient-reported outcome measure for assessment and clinical decision-making in patients with knee OA with good psychometric properties (ORNETTI et al., 2011).
Physical function | Follow up period (week 18).
  Physical function will be measured by Knee Injury and Osteoarthritis Outcome Score (KOOS) using an Activities of Daily Living subscale. The KOOS is a patient-reported outcome measure composed of 42 items divided into five subscales: Pain, other Symptoms, Activities of daily living, Sport and Recreation Function, and Knee-related Quality of Life. Its score ranges from 0 (extreme problem) to 100 (no problems) separately in each subscale (COLLINS et al., 2011). The Brazilian version of the KOOS questionnaire was recently validated, consisting of an instrument with validity, reliability, and responsiveness in patients with knee OA (ALMEIDA et al., 2022).
Pain score | Baseline (week 0), During intervention (week 6), Post-intervention (week 12), Follow up period (week 18).
  Pain will be measured by Knee Injury and Osteoarthritis Outcome Score using the pain subscale. Its score ranges from 0 (extreme problem) to 100 (no problems) (COLLINS et al., 2011).
Other Symptoms | Baseline (week 0), During intervention (week 6), Post-intervention (week 12), Follow up period (week 18).
  Other symptoms (hear clicking, swelling, catching, restricted range of motion, and stiffness) will be measured by Knee Injury and Osteoarthritis Outcome Score using the other symptoms subscale. Its score ranges from 0 (extreme problem) to 100 (no problems) (COLLINS et al., 2011).
Sport and Recreation Function | Baseline (week 0), During intervention (week 6), Post-intervention (week 12), Follow up period (week 18).
  Sport and Recreation Function will be measured by Knee Injury and Osteoarthritis Outcome Score using the Sport and Recreation Function subscale. Its score ranges from 0 (extreme problem) to 100 (no problems) (COLLINS et al., 2011).
Knee-related Quality of Life | Baseline (week 0), During intervention (week 6), Post-intervention (week 12), Follow up period (week 18).
  Knee-related Quality of Life will be measured by Knee Injury and Osteoarthritis Outcome Score using the Knee-related Quality of Life subscale. Its score ranges from 0 (extreme problem) to 100 (no problems) (COLLINS et al., 2011).
Pain catastrophizing | Baseline (week 0), During intervention (week 6), Post-intervention (week 12), Follow up period (week 18).
  Pain Catastrophizing Scale will measure pain catastrophizing. This instrument is a self-administered questionnaire, validated, translated into Brazilian Portuguese, and used to classify subjects with chronic pain as potential catastrophizers (SEHN et al., 2012; SULLIVAN, BISHOP, and PIVIK, 1995). The scale consists of 13 items related to self-reported catastrophic thoughts, feelings, and behaviors. Items are rated on a 5-point Likert scale, ranging from 0 to 4, and the total score is generated by summing the scores of all items (0-52). Higher values indicate catastrophic thoughts about pain.
Symptoms of depression, anxiety, and stress | Baseline (week 0), During intervention (week 6), Post-intervention (week 12), Follow up period (week 18).
  Symptoms of depression, anxiety, and stress will be measured by Depression, Anxiety, and Stress Scale, which is a self-reported instrument validated and translated into Brazilian Portuguese (VIGNOLA and TUCCI, 2014). It consists of 21 items ranging from 0 to 3, divided into subscales of seven questions each. The highest score on each subscale represents more significant symptoms severity of depression, anxiety, and stress.
Sleep quality | Baseline (week 0), During intervention (week 6), Post-intervention (week 12), Follow up period (week 18).
  The Pittsburgh Sleep Quality Index will measure sleep quality. The questionnaire, validated for the Brazilian population, comprises 19 self-reported questions and five questions directed to the roommate about sleeping habits in the last month. Questions directed to the roommate will not be considered as they are used to obtain clinical information. Thus, the 19 questions are categorized into seven components, graded on a score that ranges from 0 to 3. The sum of the scores of the seven components (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disorders, use of sleeping medication, and daytime dysfunction) will result in a global score (0 to 21), where the highest score indicates worst sleep quality.
Sit-to-stand activity | Baseline (week 0), and Post-intervention (week 12).
  The 30-s chair-stand test will measure sit-to-stand activity (DOBSON et al., 2013). Participants will be instructed to sit in the center of the chair, which will be positioned against the wall, with their upper limbs resting on their chest and their feet slightly apart and aligned with their hips. Initially, the participant will perform the test movements for familiarization and be instructed to sit down and get up from the chair as quickly as possible within 30 seconds. Thus, the measurement result will consist of a total number of complete chair stands in 30 s (up and down represent one stand) (Jones, Rikli, and Beam, 1999).
Ambulatory transition activity | Baseline (week 0), and Post-intervention (week 12).
  The Timed Up & Go test will measure ambulatory transition activity (DOBSON et al., 2013). Participants will be instructed to move from a seated position to standing, walk to a mark of 3 m, turn around, and return to the starting position. The measurement result will be expressed in seconds corresponding to task's completion period.
Short distance walking activity | Baseline (week 0), and Post-intervention (week 12).
  The 40 m fast-paced walk test will measure short-distance walking activity (DOBSON et al., 2013). Subjects will be instructed to walk as quickly but as safely as possible, without running at the 10 m mark, turn around, and return, then repeat for 40m. The measurement of walking time will only consist of the 10 m walking period, excluding turns. The speed measurement will be expressed in m/s, dividing the 40 m by the time (seconds) needed to travel through the test area.
Stair negotiation activity | Baseline (week 0), and Post-intervention (week 12).
  The Stair Climb Test will measure the subject's ability to climb stairs (DOBSON et al., 2013). Subjects will be instructed to ascend and descend stairs as quickly as possible using their usual shoes. The measurement will be expressed in seconds, corresponding to the total time taken for both ascending and descending the stairs.
Quadriceps femoris muscle thickness | Baseline (week 0), and Post-intervention (week 12).
  The quadriceps muscle thickness will initially be measured according to quadriceps femoris images generated by muscle ultrasound. Subsequently, this measurement will be reproduced in Image-J software (National Institutes of Health, USA, version 1.53) considering the distance between the muscle fascia or at the fascia and bone structure interface (TANIGUCHI et al., 2015). The muscle thickness will be expressed in centimeters and presented as the sum of the measurements of each quadriceps femoris muscle, with individual muscle values also shown separately
Quadriceps femoris muscle quality | Baseline (week 0), and Post-intervention (week 12).
  Quadriceps muscle quality will be expressed as quadriceps femoris muscle echo intensity generated by muscle ultrasound and measured using a specific function (greyscale) in Image J software. The echo intensity value of the region of interest will be expressed in arbitrary units, ranging between 0 (black) and 255 (white) (PARIS e MOURTZAKIS, 2021). The highest value represents decreased muscle quality and deposition of non-contractile tissue within the muscle. The echo intensity data will be corrected according to subcutaneous fat thickness. Data will be presented as the mean of the echogenicity of the quadriceps femoris, with individual muscle values also shown separately.
Pennation angle | Baseline (week 0), and Post-intervention (week 12).
  Measurement of the pennation angle will be performed using only images of the vastus lateralis due to the alignment of the fascicles (BLAZEVICH et al., 2007). The pennation angle is formed between the muscle fascicle line and the deep aponeurosis. It will be expressed in degrees. The mean of three measurements for pennation angle will be presented.
Fascicle length | Baseline (week 0), and Post-intervention (week 12).
  Measurement of the fascicle length will be performed using only images of the vastus lateralis due to the alignment of the fascicles (BLAZEVICH et al., 2007). Fascicle length is characterized by the distance of the fascicle between the superficial and deep aponeurosis. It will be estimated (in cm) from muscle thickness and fascicle pennation angle using a padronized equation. The mean of three measurements for fascicle angle will be presented.

OTHER OUTCOMES:
Number of medications | Baseline (week 0), During intervention (week 6), Post-intervention (week 12), Follow up period (week 18).
  The number of analgesic and anti-inflammatory medications ingested will be measured considering information reported by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Cristine Lima Alberton, PhD, Principal Investigator — Federal University of Pelotas
Locations (1):
- Federal University of Pelotas, Pelotas, Brazil, Pelotas, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ornetti P, Dougados M, Paternotte S, Logeart I, Gossec L. Validation of a numerical rating scale to assess functional impairment in hip and knee osteoarthritis: comparison with the WOMAC function scale. Ann Rheum Dis. 2011 May;70(5):740-6. doi: 10.1136/ard.2010.135483. Epub 2010 Dec 13. PMID 21149497
- [Background] Collins NJ, Misra D, Felson DT, Crossley KM, Roos EM. Measures of knee function: International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form, Knee Injury and Osteoarthritis Outcome Score (KOOS), Knee Injury and Osteoarthritis Outcome Score Physical Function Short Form (KOOS-PS), Knee Outcome Survey Activities of Daily Living Scale (KOS-ADL), Lysholm Knee Scoring Scale, Oxford Knee Score (OKS), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), Activity Rating Scale (ARS), and Tegner Activity Score (TAS). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S208-28. doi: 10.1002/acr.20632. No abstract available. PMID 22588746
- [Background] Almeida GPL, da Costa RMO, Albano TR, Tavares MLA, Marques AP. Translation, cross-cultural adaptation, validation and responsiveness in the Brazilian Portuguese version of the Knee Injury and Osteoarthritis Outcome Score (KOOS-BR). Knee Surg Sports Traumatol Arthrosc. 2022 Oct;30(10):3343-3349. doi: 10.1007/s00167-022-06911-w. Epub 2022 Feb 26. PMID 35218377
- [Background] Sehn F, Chachamovich E, Vidor LP, Dall-Agnol L, de Souza IC, Torres IL, Fregni F, Caumo W. Cross-cultural adaptation and validation of the Brazilian Portuguese version of the pain catastrophizing scale. Pain Med. 2012 Nov;13(11):1425-35. doi: 10.1111/j.1526-4637.2012.01492.x. Epub 2012 Oct 4. PMID 23036076
- [Background] Vignola RC, Tucci AM. Adaptation and validation of the depression, anxiety and stress scale (DASS) to Brazilian Portuguese. J Affect Disord. 2014 Feb;155:104-9. doi: 10.1016/j.jad.2013.10.031. Epub 2013 Oct 28. PMID 24238871
- [Background] Bertolazi AN, Fagondes SC, Hoff LS, Dartora EG, Miozzo IC, de Barba ME, Barreto SS. Validation of the Brazilian Portuguese version of the Pittsburgh Sleep Quality Index. Sleep Med. 2011 Jan;12(1):70-5. doi: 10.1016/j.sleep.2010.04.020. Epub 2010 Dec 9. PMID 21145786
- [Background] Dobson F, Hinman RS, Roos EM, Abbott JH, Stratford P, Davis AM, Buchbinder R, Snyder-Mackler L, Henrotin Y, Thumboo J, Hansen P, Bennell KL. OARSI recommended performance-based tests to assess physical function in people diagnosed with hip or knee osteoarthritis. Osteoarthritis Cartilage. 2013 Aug;21(8):1042-52. doi: 10.1016/j.joca.2013.05.002. Epub 2013 May 13. PMID 23680877
- [Background] Jones CJ, Rikli RE, Beam WC. A 30-s chair-stand test as a measure of lower body strength in community-residing older adults. Res Q Exerc Sport. 1999 Jun;70(2):113-9. doi: 10.1080/02701367.1999.10608028. PMID 10380242
- [Background] Taniguchi M, Fukumoto Y, Kobayashi M, Kawasaki T, Maegawa S, Ibuki S, Ichihashi N. Quantity and Quality of the Lower Extremity Muscles in Women with Knee Osteoarthritis. Ultrasound Med Biol. 2015 Oct;41(10):2567-74. doi: 10.1016/j.ultrasmedbio.2015.05.014. Epub 2015 Jun 20. PMID 26099784
- [Background] Paris MT, Mourtzakis M. Muscle Composition Analysis of Ultrasound Images: A Narrative Review of Texture Analysis. Ultrasound Med Biol. 2021 Apr;47(4):880-895. doi: 10.1016/j.ultrasmedbio.2020.12.012. Epub 2021 Jan 13. PMID 33451817
- [Background] Blazevich AJ, Cannavan D, Coleman DR, Horne S. Influence of concentric and eccentric resistance training on architectural adaptation in human quadriceps muscles. J Appl Physiol (1985). 2007 Nov;103(5):1565-75. doi: 10.1152/japplphysiol.00578.2007. Epub 2007 Aug 23. PMID 17717119
- [Derived] Carvalho MTX, Alberton CL. Remote and In-person Supervised Exercise in Patients with Knee Osteoarthritis (RISE-KOA): study protocol for a non-inferiority randomized controlled trial. Trials. 2025 May 20;26(1):165. doi: 10.1186/s13063-025-08884-w. PMID 40394687